CLINICAL TRIAL: NCT05079347
Title: Traditional Healer-initiated HIV Counseling and Testing in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carolyn Audet, Assistant Professor of Preventive Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201977; 1R34MH124496-01A1 (NIH)
Record Dates: First submitted 2021-10-01; First posted 2021-10-15 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: HIV Infection
Keywords: HIV testing; HIV stigma; Trust in health care provider
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: We will pilot the intervention with a small group of traditional healers who will offer HIV testing to their patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healer led HIV testing (Experimental): Traditional healers will offer HIV testing to their patients. They will provide the test result to patients. If the patient is positive they will refer their patients to the health facility via referral form and/or walk them to the clinic (based on patient preference). If the patient is negative, the healer will encourage them to re-test at the health facility in 6 months during an "open house" event where healers will attend to try and de-stigmatize going to the health facility.
  Interventions: Diagnostic Test: HIV rapid test

INTERVENTIONS:
Diagnostic Test: HIV rapid test — Using a rapid test to assess a patient's HIV status

SUMMARY:
The objective of this proposal is to conduct a pilot test of a program aimed at training traditional healers to conduct HIV testing and implementing HIV testing among people living in Bushbuckridge, South Africa.

Pilot Healer-initiated HIV testing uptake and linkage to prevention services. Trust in allopathic health care and HIV stigma will be measured among participants at study enrollment and at month seven.

Hypothesis: Healer-initiated HIV counseling and testing (HICT) will increase trust in allopathic health care and reduce HIV stigma.

DETAILED DESCRIPTION:
Traditional healers see patients who avoid allopathic health services, including those who refuse HIV testing. Patients report a general preference for traditional healers, given their fluency in local language, the length of time they spend with patients, the respect they show patients, the cultural congruity to their diagnosis, and their proximity to the patients. Reports of poor treatment by health care providers are common in SSA, often resulting in patients refusing or delaying allopathic health services and/or seeking alternative health services. Men, immigrants, and those with low SES most frequently report poor treatment at the health facility or report that the health system is not designed for their needs. People who first visit a traditional healer for HIV-associated symptoms before seeking an HIV test are delayed 2.4 times longer in seeking health services than those who do not. Among patients enrolled in HIV care and treatment, a preference for traditional medicine impacts their treatment decisions: patients who report use of both traditional and allopathic services are 45% less likely to enroll in antiretroviral therapy (ART) services.

Healers are respected members of their communities, play an integral role as informal referral agents to the South African health system, and act as supportive providers to patients living with chronic disease, if effectively engaged. In rural South Africa, traditional healers provide physical and psychological services to >80% of the population. There are more than 200,000 traditional healers in South Africa, but only 46,000 registered physicians (> 20:1 ratio) who provide services for a myriad of disease conditions, including HIV, TB, malaria, epilepsy, schizophrenia, and depression. Given the level of trust in the community and the numbers of healers, partnerships may facilitate diagnosis and linkage to care via the creation of unique testing locations. It is up to researchers and health care providers to overcome our own biases and/or prejudices against this workforce to develop an effective strategy to increase testing uptake.

Traditional healers can bridge the testing gap between "non-testers" and the allopathic health system. Traditional healers have been successfully engaged in health systems to promote care linkage among people living with diabetes, TB, HIV, malaria, and mental illness- many of whom initially did not believe in their allopathic diagnosis until a healer convinced them that their condition was not caused by a curse. Those who are hesitant to test need a trusted and culturally concordant provider (traditional healer) to both vouch for and deliver the HIV test, and the same provider to create a bridge to the allopathic health facility, providing a metaphorical "safe space" for the patient while they transition to HIV care. Traditional healers are strongly motivated to play this role for two reasons: (1) Better patient health outcomes are strongly correlated with perceived quality of traditional healer care. Healers do not want to be associated with high levels of morbidity or mortality, as it is bad for business; and (2) Healers are excited at expanding their public health services. As allopathic medical knowledge is disseminated, healer views on disease causation are expanding to include the germ theory of disease. Patients are open to this partnership, given their inclination to ping-pong between the two systems depending on their needs.

ELIGIBILITY:
Inclusion Criteria:

1. Traditional healers > 18 years of age, who are registered as traditional healers with the government of South Africa, are currently practicing in the Bushbuckridge area, and are trained to provide HIV testing.
2. Biomedical practitioners > 18 years of age, who are currently providing HIV-related health care services to patients at government or private health facilities in Bushbuckridge.
3. Community members > 18 years of age, who have not received an HIV test result in the past year and who currently live in Bushbuckridge.

Exclusion Criteria:

1. Traditional healers who do not believe in HIV disease and those who can not pass their HIV counseling and testing certification.
2. Biomedical practitioners who do not interact with patients seeking treatment for HIV.
3. Community members who are not out sound mind or body during the recruitment (inebriated, too sick to leave the house) and community members with a previous positive HIV test result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Audet, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Thulamahashe Health Facility, Thulamahashi, Mpumalanga, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of healer clients took place between July 22, 2022, to May 31, 2023, at the homes of the traditional healers. Healers were not recruited as they were considered employed by the study.
Pre-assignment Details: We only recruited and enrolled the clients of traditional healers. The healers themselves were not considered enrolled. Those who self-reported a positive HIV test were excluded from the study.
  Those enrolled were offered HIV testing by the healer. We looked at the uptake of testing; so we have demographic data on those who enrolled (n= 418) but not on those who refused (n=93) or those who self reported being HIV+ (n=64).
Period: Overall Study
Arm/Group | Healer Led HIV Testing
Started (418 people said they would be interested in receiving an HIV test from the healer) | 418
Completed (418 people actually went through with the test and received their results) | 418
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healer Led HIV Testing
Number analyzed (Participants) | 418
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214
  Male | 204
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 418
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 418

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Completing HIV Testing Training
Description: Percentage of healers who are able to complete the training program.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Healer Led HIV Testing
Number analyzed (Participants) | 17
Participants | 16

2. Primary Outcome: Uptake of HIV Testing
Description: the percentage of people who are accept testing/ approached to complete testing
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Healer Led HIV Testing
Number analyzed (Participants) | 418
Participants | 418

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Healer Led HIV Testing
All-Cause Mortality (participants affected / at risk) | 0/418
Serious Adverse Events (participants affected / at risk) | 0/418
Other Adverse Events (participants affected / at risk) | 0/418

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT05079347/Prot_SAP_001.pdf
  • Informed Consent Form (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT05079347/ICF_000.pdf